CLINICAL TRIAL: NCT01949974
Title: Integral Attention Program With or Without Palliative Chemotherapy in Advanced Cancer Patients: A Randomized Multicenter Clinical Trial
Brief Title: Integral Attention Program With or Without Palliative Chemotherapy in Advanced Cancer Patients
Acronym: PAI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Dificulties in the recruitment of patients.
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIBSP-PAI-2011-36; 2012-001128-36 (EudraCT Number); PI11/01366 (Other Grant/Funding Number: Institute of Health Carlos III)
Record Dates: First submitted 2013-09-17; First posted 2013-09-25 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2013-08

CONDITIONS: Cancer
Keywords: Palliative Chemotherapy; Integral Attention Program; Advanced cancer; Randomized Clinical Trial
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integral Attention Program (PAI) (Experimental): The key points of the PAI are:
  * To assess and manage pain and other symptoms resulting from disease progression.
  * To evaluate the information needs that may arise and to address them.
  * To encourage patient and family adaptation to the situation of advanced disease and in the terminal phase of it.
  * To provide guidance in decision-making while respecting patient autonomy.
  * To establish a plan of care and treatment, adapted to the evolution and needs of the patient.
  * To promote continuity of care.
  Interventions: Other: Integral Attention Program (PAI)
- Standard Palliative Chemotherapy and PAI (Active Comparator): Standard palliative chemotherapy will be administered, depending on type of cancer, as well as PAI as been defined above.
  Interventions: Drug: Standard Palliative Chemotherapy; Other: Integral Attention Program (PAI)

INTERVENTIONS:
Drug: Standard Palliative Chemotherapy — Standard Palliative Chemotherapy, depending on type cancer.
  Arms: Standard Palliative Chemotherapy and PAI
Other: Integral Attention Program (PAI) — The PAI is a plan of care and treatment adapted in accordance with the evolution and needs of patients. This plan includes an initial comprehensive assessment of patients and their families during the first visit, including specialized psychological and social support when needed, voluntary art therapy and/or mindfulness. There will be outpatient monitoring, 24h phone assistance, home visits, support should hospitalization be required, and unscheduled visits by a palliative care team.

SUMMARY:
The purpose of this clinical trial is to compare a non-pharmaceutical intervention (Integral Attention Program or PAI) versus standard palliative chemotherapy treatment plus PAI in patients with advanced cancer who have already received at least a first course of chemotherapy but had proven therapeutic failure.

The study hypothesis is that palliative chemotherapy offers no clear benefits in relation to quality-of-life-adjusted survival compared to a comprehensive care program.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age.
* Patients potentially eligible to receive a new chemotherapy cycle and whose clinical condition, according to the oncologist, does not identify any therapeutic strategy clearly superior to another, in the light of scientific evidence.
* Patients with advanced cancers that have been treated with chemotherapy but who have not displayed complete response to treatment or who, after treatment response, are now in a situation of recurrence or disease progression
* Patients who have previously received at least one chemotherapy cycle of the following tumors:

  * Cancer of the digestive and gastrointestinal tract
  * Head and Neck Cancer
  * Lung cancer
  * Urologic cancers
  * Gynecologic cancers
  * Central nervous system cancer
  * Melanoma
* Patients who can potentially comply with study and/or monitoring procedures and to accept and sign the informed consent form.
* Patients whose home is located less than 10 km, approximately, of the hospitals participating in the study.

Exclusion Criteria:

* Patients who are currently receiving chemotherapy, although patient pursuing any other concomitant treatment are eligible (eg, hormone therapy or radiation therapy).
* Patients who have contraindications to chemotherapy.
* Patients who did not agree to participate in the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Survival adjusted for quality of life | At one year of follow-up
  Quality of life will be measured by the EuroQoL-5D questionnaire.

SECONDARY OUTCOMES:
Specific Quality of life: measured through the quality of life questionnaire of the European Organisation for Research and Treatment of Cancer (EORTC QLQ C-30) and Palliative Care Scale (POS) | At one year of follow-up
Control of symptoms using the Edmonton Symptom Assessment System | At one year of follow-up
Toxicity by the American National Cancer Institute toxicity | At one year of follow-up
Patient satisfaction regarding care using a Likert scale of 5 items (very satisfied, satisfied, neither satisfied or dissatisfied, somewhat satisfied and not satisfied). | At one year of follow-up
Costs reported by the information system of each hospital | At the end of follow-up
Adverse effects related to study interventions | At one year of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pascual, Dr., PhD, Principal Investigator — Palliative Unit. Clinical Oncology Service. Hospital de la Santa Creu i Sant Pau. Barcelona. Spain.
Locations (3):
- Spain (3):
  - Hospital General de l'Hospitalet de Llobregat, L'Hospitalet de Llobregat, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona